CLINICAL TRIAL: NCT04303741
Title: An Open-labeled, Single-arm, Investigator-initiated Phase II Trial of Camrelizumab (Anti-PD-1 Antibody) in Combination With Apatinib and Eribulin in Patients With Advanced Triple-Negative Breast Cancer
Brief Title: A Phase II Trial of Camrelizumab in Combination With Apatinib and Eribulin in Patients With Advanced TNBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immuno2020-01
Record Dates: First submitted 2020-03-07; First posted 2020-03-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; apatinib; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab +Apatinib+Eribulin (Experimental): Camrelizumab 200mg(3mg/kg for patient whose weight is below 50kg) iv Q3W combination with Apatinib 250mg, po, daily (d1-d21)and Eribulin1.4mg/m2 iv d1, d8 Q3W
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Drug: Eribulin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg (3mg/kg for patient whose weight is below 50kg) will be administered as an intravenous infusion over 30 minutes every three weeks until unacceptable toxic effects or disease progression or other termination criteria appeared. Patients received up to two years of treatment.
Drug: Apatinib — Apatinib 250mg will be administered daily until unacceptable toxic effects or disease progression or other termination criteria appeared. Patients received up to two years of treatment.
Drug: Eribulin — Eribulin Mesylate will be administered as a 1.4 mg/m2 intravenous (IV) injection over 2 to 5 minutes on day 1 and day 8 of each 21-day cycle until unacceptable toxic effects or disease progression or other termination criteria appeared. Patients received up to two years of treatment.
  Other Names: Eribulin Mesylate

SUMMARY:
This is a phase II, open-labeled, multi-centered,single-arm, Investigator-initiated clinical trial of camrelizumab (an anti-PD-1 antibody) in combination with apatinib (a VEGFR2 TKI) and eribulin mesylate in patients with advanced triple-negative breast cancer. We will enroll 46 subjects (Simons two stage design). This study aims to evaluate the efficacy and safety of camrelizumab combined with apatinib and eribulin in the treatment of advanced TNBC.

DETAILED DESCRIPTION:
This a phase II, open-labeled, multi-centered, single-arm, investigator-initiated clinical trial to assess the efficacy and safety of camrelizumab combination with apatinib and eribulin in female patients age of 18 to 70 with advanced TNBC, and previously treated with at least one line of systemic therapy in the advanced setting. Prior therapy (adjuvant/neoadjuvant/advanced) must have included an anthracycline and a taxane. The number of patients to be included is 46 patients (Simons two stage design). The primary objective is to assess the overall response rate (ORR). All enrolled patients will be treated with camrelizumab 200mg (iv. 3mg/kg for patient whose weight is below 50kg) on day 1 of each 21-day cycle, and apatinib 250mg daily (po, d1-d21), in combination with eribulin mesylate at 1.4 mg/m2 (iv.) on day 1 and day 8 of every 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. The patients sign the written informed consent.
2. Women aged 18-70.
3. The pathologic diagnosis of unresectable recurrent or metastatic triple-negative breast cancer ［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］. Patients with at least one measuring lesion that was conformed to RECIST v1.1 standard.
4. Prior therapy (adjuvant/neoadjuvant/advanced) must have included an anthracycline and a taxane in any combination or order and either in the early or metastatic disease setting unless contraindicated for a given patient.
5. The patient can swallow pills.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. With a life expectancy of at least 12 weeks.
8. The results of patient's blood tests are as follows:

   • Hb≥90g/L; • Plt≥100^9/L; • Serum albumin ≥3g/dL;• Neutrophils≥1.5^9/L; TSH≤ normal upper limit (ULN);• ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN); • TBIL ≤ULN (total bilirubin ≤1.5 ULN in Gilbert's syndrome or liver metastasis subjects);• ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN);• AKP≤ 2.5 ULN; • Renal function within 7 days before the first administration: serum creatinine ≤1.5 ULN or creatinine clearance ≥60mL/min
9. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 6 months after the last dose of study treatment.

Exclusion Criteria:

1. The subjects had a central nervous system metastases with clinical symptoms.
2. Other clinical trials of drugs were used in the first four weeks before the first dose.
3. Subjects with severe allergic reactions to other monoclonal antibodies.
4. Received other anti-tumor treatments within 28 days before the first dose.
5. A heart condition or disease that is not well controlled.
6. Subjects with treatment history of anti-angiogenesis drugs, or immunotherapy (previous use of anti-PD-1/PD-L1 antibodies was allowed) or eribulin.
7. The subjects had any history of autoimmune disease or any use of systemic glucocorticoid or immunosuppressive medications.
8. Subjects had history of hypertension and poor control with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
9. Urine routine indicated that urine protein ≥ ++, or the 24-hour urine protein quantity ≥ 1.0g.
10. Hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.).
11. Congenital or acquired immune deficiency (such as HIV infection);
12. Receive live vaccine within 4 weeks before or during the study period;
13. Patients who are allergic to or contraindicated to the experimental drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | from the first drug administration up to the first occurrence of progression or death (up to 24 months)
  The propotion of subjects with CR or PR.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from the first drug administration to within 90 days for the last dose
  Adverse events/serious adverse events
Disease Control Rate (DCR) | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  The propotion of subjects with CR, PR, or SD.
DOR | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  Duration of response
PFS | from the first drug administration up to the first occurrence of progression or death (up to 24 months)
  Progression-Free-Survival
One year-OS rate | 12 months after the first drug administration
  One year-Overall survival rate
Clinical benefit rate (CBR) | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  The propotion of subjects with CR, PR, or SD for >=6 months during the study.
TTR | from the first drug administration up to one year
  Time to response
Frequencies of Biomarkers | pre-treatment, up to 24 months
  Biomarkers (including tumor/stromal PD-L1, stromal PD-1, tumor-infiltrating lymphocytes and tumor-infiltrating B cells, eg)

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Changhai Hospital, Navy Medical University (Second Military Medical University), Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Wang Y, Tian Z, Lin Y, Li H, Zhu Z, Liu Q, Su S, Zeng Y, Jia W, Yang Y, Xu S, Yao H, Jiang W, Song E. Multicenter phase II trial of Camrelizumab combined with Apatinib and Eribulin in heavily pretreated patients with advanced triple-negative breast cancer. Nat Commun. 2022 May 31;13(1):3011. doi: 10.1038/s41467-022-30569-0. PMID 35641481